CLINICAL TRIAL: NCT00208663
Title: Validation of an Instrument to Qualitatively and Quantitatively Profile Hospitalist Workflow
Status: Withdrawn | Type: Observational
Why Stopped: Resources
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Jason Stein, MD, Assistant Professor, Emory University
Other Study IDs: 814-2005
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: Physician Workflow

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine if a simple 'pick-list' menu applied to a handheld computer's time-motion program can be used to record reliably what a hospital-based doctor does while working a shift in the hospital. In this study reliability will be measured by comparing the data collected by at least two different observers recording data from the same hospitalist during the same period of time.

DETAILED DESCRIPTION:
We were unable to configure the software to get started on this study.

ELIGIBILITY:
Inclusion Criteria:

* Must be a practicing hospitalist, defined as a physician working exclusively in a hospital settings

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Physicians
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2005-09; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Elapsed time engaged in specific hospital work activities | 1 hospital workday

CONTACTS AND LOCATIONS:
Overall Officials: Jason M Stein, MD, Principal Investigator — Emory University
Locations (1):
- Emory affiliated hospitals, Atlanta, Georgia, United States

REFERENCES:
- [Background] Gillanders W, Heiman M. Time study comparisons of 3 intern programs. J Med Educ. 1971 Feb;46(2):142-9. doi: 10.1097/00001888-197102000-00005. No abstract available. PMID 5540257
- [Background] Lurie N, Rank B, Parenti C, Woolley T, Snoke W. How do house officers spend their nights? A time study of internal medicine house staff on call. N Engl J Med. 1989 Jun 22;320(25):1673-7. doi: 10.1056/NEJM198906223202507. PMID 2725617
- [Background] Parenti C, Lurie N. Are things different in the light of day? A time study of internal medicine house staff days. Am J Med. 1993 Jun;94(6):654-8. doi: 10.1016/0002-9343(93)90220-j. PMID 8506894
- [Background] PAYSON HE, GAENSLEN EC Jr, STARGARDTER FL. Time study of an internship on a university medical service. N Engl J Med. 1961 Mar 2;264:439-43. doi: 10.1056/NEJM196103022640906. No abstract available. PMID 13733711